CLINICAL TRIAL: NCT01198730
Title: Screen of Diabetes Mellitus by Oral Glucose Tolerance Test in Subjects Receiving Catheterization or Multi-detector Computed Tomography (MDCT) for Coronary Artery Disease
Brief Title: Screen of DM by OGTT in Subjects Receiving CAG or MDCT for CAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Chief in Internal medicine department, Taichung Veterans General Hospital
Other Study IDs: C08215
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
Keywords: DM; CAD; Meal tolerance test
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected during OGTT after an overnight fasting
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the glucose regulation status of patients who were suspected to have CAD in central Taiwan.

DETAILED DESCRIPTION:
It had been reported that high prevalence of IGT (impaired glucose tolerance) and unknown DM (diabetes mellitus) in patients with CAD (coronary artery disease). This study aimed to determine the glucose regulation status of patients who were suspected to have CAD in central Taiwan. In general, patient who were admitted for CAG (coronary angiography) or MDCT without known DM were eligible. After informed consent, OGTT (oral glucose tolerance test) was performed to determine the glucose regulation status. Study participants will be requested to complete questionnaires to assess their risk of diabetes and quality of sleep. Patients who were diagnosed as new DM would be asked to follow up in clinical service with diet control.

ELIGIBILITY:
Inclusion Criteria:

* Patient received CAG or MDCT for suspect CAD
* Without DM history

Exclusion Criteria:

* Known DM
* Unstable disease condition
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study, we screened adult patients admitted for coronary angiography due to angina
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diabetes | 3 months
  Based on OGTT and HbA1c

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor | 3 months
  An biomarker to link brain and atheroclerosis
Coroanry artery disease | 3 months
  Based on coronary angiography and medical record
Mortality | 5 years
  All-cause and cardiovascular

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H-H Sheu, MD, PHD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Liang KW, Lee WJ, Lee IT, Lee WL, Wang JS, Wu JP, Sheu WH. Subjects with microvascular angina have longer GT repeats polymorphism in the haem oxygenase-1 gene promoter. Biomarkers. 2020 Mar;25(2):144-148. doi: 10.1080/1354750X.2020.1713214. Epub 2020 Jan 20. PMID 31916865
- [Derived] Liang KW, Sheu WH, Lee WJ, Lee WL, Fu CP, Wang JS. Differential expression of circulating vascular cell adhesion molecule-1 in subjects with coronary artery disease and cardiac syndrome X without known diabetes mellitus. Biomarkers. 2017 Dec;22(8):798-804. doi: 10.1080/1354750X.2017.1351003. Epub 2017 Jul 18. PMID 28675064
- [Derived] Liang KW, Sheu WH, Lee WJ, Lee WL, Pan HC, Lee IT, Wang JS. Post-challenge insulin concentration is useful for differentiating between coronary artery disease and cardiac syndrome X in subjects without known diabetes mellitus. Diabetol Metab Syndr. 2017 Feb 8;9:10. doi: 10.1186/s13098-017-0209-1. eCollection 2017. PMID 28194232
- [Derived] Wang JS, Lee IT, Lee WJ, Lin SY, Fu CP, Ting CT, Lee WL, Liang KW, Sheu WH. Performance of HbA1c and fasting plasma glucose in screening for diabetes in patients undergoing coronary angiography. Diabetes Care. 2013 May;36(5):1138-40. doi: 10.2337/dc12-1434. Epub 2012 Dec 13. PMID 23238660